CLINICAL TRIAL: NCT04805398
Title: A Randomized, Double Blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy, Safety, PK, PD and Immunogenicity of Subcutaneously Given Multiple-Dose CM310 in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: Subcutaneously CM310/Placebo in Patients With Chronic Rhinosinusitis With Nasal Polyposis (CROWNS-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310NP001
Record Dates: First submitted 2021-03-12; First posted 2021-03-18 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2021-11

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Nasal Polyps
Keywords: Chronic Rhinosinusitis with Nasal Polyps
MeSH Terms: conditions — Disease; Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 (Experimental): CM310 300mg is given subcutaneously (SC) every two weeks for 16-week treatment
  Interventions: Biological: CM310
- Placebo (Placebo Comparator): Placebo is given subcutaneously (SC) every two weeks for 16-week treatment.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CM310 — 300 mg every two weeks
  Arms: CM310
Biological: Placebo — 300 mg every two weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled study to evaluate the efficacy, safety, PK, PD and immumogenicity of CM310 in comparison to placebo in addition to a background treatment of mometasone furcate nasal spray (MFNS) in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP).

DETAILED DESCRIPTION:
The study consists of a Screening/run-in Period (up to 4 weeks), a Randomized, Double Blind Treatment Period (16 weeks, till End-of-Treatment Visit) and a Safety Follow-up Period (8 weeks, till End-of-Study Visit).

56 patients who meet eligibility criteria will be randomized 1:1 to receive either CM310 300mg or matched placebo subcutaneously every two weeks (Q2W) for a total of 8 times. All patients will receive MFNS on a daily basis as a background treatment throughout the study. MFNS is required to use no less than 14 days during Screening/run-in Period.

Central reading will be implemented to nasal endoscopic nasal polyp score (NPS) , CT scans to Lund-Mackay score and volume of the involved area of nasosinusitis on 3D-construction images, and nasal polyp biopsy tissue analysis to eosinophil counts & percentage.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral CRSwNP.
* Prior treatment with systemic corticosteroids (SCS), and/or contraindicate to or intolerance to SCS, and/or with prior surgery to nasal polyps.
* Stable dose of intranasal corticosteroids for at least 4 weeks before screening.
* Ongoing symptoms for at least 4 weeks before screening：1)Nasal congestion/obstruction; 2)Othe symptom, e.g., loss of smell or rhinorrhea.
* Bilateral NPS of ≥5 with a minimum score of 2 in each nasal cavity at screening and at baseline.
* NCS score of 2 or 3 at screening and at baseline.
* Eosinophilic level meets the one of the following criteria: 1) serum eosinophil count ≥6.9% (without concomitant asthma) or ≥3.7% (with concomitant asthma) at screening; 2) absolute count of ≥55 per high power field or percentage of ≥27% in eosinophil level from nasal polyps biospy tissue.
* Contraception.

Exclusion Criteria:

* Not enough washingout period for previous therapy, e.g., less than 10 weeks or 5 half-lives (whichever is longer) for IL-4Rα antagonists, less than 8 weeks or 5 half-lives for biologic therapy/systemic immunosuppressant, less than 6 months for sinus surgery (including polypectomy).
* concurrent disease, e.g., ongoing rhinitis medicamentosa, acute sinusitis, nasal infection or upper respiratory infection, allergic fungal rhinosinusitis, malignancy, uncontrolled chronic disease such as cardivascular diseases, tuberculosis, diabetes etc.
* Allergic or intolerant to mometasone furoate spray or CM310/placebo.
* Significant liver or renal dysfunction.
* Other.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Bilateral endoscopic Nasal Polyps Score (NPS) | at Week 16
  Change from baseline in the bilateral endoscopic NPS.NPS score ranges from 0-8. (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Nasal Congestion/Obstruction SymptomSeverity (NCS) Score | at Week 16
  Change from baseline in the NCS score. NCS score (0-3), higher score means worse nasal symptom.

SECONDARY OUTCOMES:
Time to the first response of NPS | Baseline up to Week 24
  Time to the first response of NPS (defined as bilateral endoscopic NPS improved ≥1).
Lund-Mackay score | at Week 16
  Change from baseline in the Lund-Mackay score on CT scan. The range of LM score is 0-24. Higher score means worse nasosinusitis.
Volume of the involved area of nasosinusitis on 3D-construction CT scan | at Week 16
  Change from baseline in the volume of the involved area of nasosinusitis on 3D-construction CT scan.
Bilateral endoscopic NPS | at Week 8
  Change from baseline in the bilateral endoscopic NPS.
Proportion of subjects receiving rescue therapy for nasal polyps | Baseline up to Week 24
  Proportion of subjects receiving rescue therapy for nasal polyps.
University of Pennsylvania Smell Identification Test (UPSIT) | at Week 16
  Change from baseline in UPSIT. UPSIT score (0-40). Higher score means better sense of smell.
22-item Sino-nasal Outcome Test Scores(SNOT-22) score | at Week 16
  Change from baseline in SNOT-22 score. SNOT-22 score (0-110). Higher score means a worse outcome.
Total Symptom Score(TSS) score | at Week 16
  Change from baseline in TSS score. TSS score (0-9). Higher score means worse nasal symptom.
Bilateral endoscopic NPS | at Week 16
  Change from baseline in the bilateral endoscopic NPS in subjects with concurrent asthma.
Bilateral endoscopic NCS | at Week 16
  Change from baseline in the NCS in subjects with concurrent asthma.
Safety parameters | Baseline up to Week 24
  Incidence of treatment-emergent adverse events (TEAEs), of treatment-emergent serious AEs (TESAEs), etc.
Pharmacokinetics(PK) | Baseline up to Week 24
  Trough concentration and exposure.
Pharmacodynamics(PD) | Baseline up to Week 24
  Change from baseline in serum biomarker level (TARC, total IgE and eosinophil level).
PD(eosinophil level in nasal polyps biospy tissue) | at Week 16
  Change from baseline of eosinophil level in nasal polyps biospy tissue.
Anti-drug antibodies(ADA) | Baseline up to Week 24
  Incidence of ADA.
Neutralizing antibody (Nab) | Baseline up to Week 24
  Incidence of Nab.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital, CMU
Locations (19):
- China (19):
  - Beijing Chaoyang Hospital, CMU, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Renmin Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shandong Second Provincial General Hospital (Shandong ENT hospital), Jinan, Shangdong
  - Renji Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Yan B, Shen S, Song X, Jiang Y, Shi L, Zhao C, Yang Y, Jiang L, Li J, Ye J, Liu J, Wan L, Yang Y, Chen J, Liu F, Su L, Xu Y, Tan G, Yu S, Zhang Y, Wang L, Liu S, Yan H, Liu W, Chen B, Wang C, Zhang L. Efficacy and safety of CM310 in severe eosinophilic chronic rhinosinusitis with nasal polyps (CROWNS-1): a multicentre, randomised, double-blind, placebo-controlled phase 2 clinical trial. EClinicalMedicine. 2023 Jul 5;61:102076. doi: 10.1016/j.eclinm.2023.102076. eCollection 2023 Jul. PMID 37483544